CLINICAL TRIAL: NCT06181942
Title: A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Urological Surgeries
Acronym: SPiM-RWS-URO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Danfeng Xu, Pro.Danfeng Xu, Ruijin Hospital
Other Study IDs: ISFMT-SP-001
Record Dates: First submitted 2023-08-17; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Urological Surgeries
Keywords: SP single-port robot; radical prostatectomy; partial nephrectomy; radical nephrectomy; radical resection of the renal pelvic carcinoma (one position); pyeloplasty and other single-port urological surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- single-port urological surgeries with the SP single-port robot: who have received or plan to receive radical prostatectomy (RP), partial nephrectomy (PN), radical nephrectomy (RN), radical resection of the renal pelvic carcinoma (one position), pyeloplasty and other single-port urological surgeries with the SP single-port robot.
  Interventions: Device: SP

INTERVENTIONS:
Device: SP — English name: da Vinci SP Surgical System Model and specification: SP1098 Manufacturer: Intuitive Surgical, Inc.

SUMMARY:
Study name：A Real-World Study to Evaluate the Clinical Performance and Safety of da Vinci SP Surgical System for Single-Port Urological Surgeries；

Study purpose：This clinical trial is a real-world study to evaluate the clinical performance and safety of da Vinci SP Surgical System ("SP single-port robot" for short) for single-port urological robotic surgeries in the real world, providing a real world evidence for clinical application of the product in the Chinese population.

Study design：Retrospective + prospective, real-world study

Investigational medical device： English name: da Vinci SP Surgical System Model and specification: SP1098 Manufacturer: Intuitive Surgical, Inc.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all the following criteria:

1. Subjects who have received or plan to receive RP, PN, RN, radical resection of the renal pelvic carcinoma (one position), pyeloplasty and other single-port urological robotic surgeries with the SP single-port robot;
2. Patients who voluntarily decide to participate in the study and sign the ICF (or exempt from signature of the ICF as approved by the EC).

Exclusion Criteria:

The subjects meeting any of the following criteria should be excluded.

1. Patients with missing data on the primary endpoint in retrospective cases;
2. Subjects having any contraindications of single-port robot surgery;
3. The intraoperative anatomy determined that minimally invasive surgery was not suitable;
4. Patients who are considered inappropriate to participate in this Study by investigators.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received or plan to receive radical prostatectomy (RP), partial nephrectomy (PN), radical nephrectomy (RN), radical resection of the renal pelvic carcinoma (one position), pyeloplasty and other single-port urological surgeries with the SP single-port robot.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative conversion rate | Intraoperative
incidence of device-related or likely related complications | 30 days

SECONDARY OUTCOMES:
Intraoperative bleeding volume | Intraoperative
The rate of intraoperative blood transfusion | Intraoperative
Surgical duration | Intraoperative
Length of stay (LOS) | up to 4 weeks
Admission to ICU and ICU LOS | up to 4 weeks
Urethral catheter indwelling duration | up to 4 weeks
Postoperative pain score | follow-ups 1 day (24±4 hours), 3 days (72±4 hours) and 1 month (30±5 days) after the surgery.
Short-term recovery of functions for1 )Erectile function and 2)Urinary continence function | in the follow-up 1 month after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided